CLINICAL TRIAL: NCT02197858
Title: Clinical Comparison of Hemodynamic Parameters Using Invasive Versus Non-invasive Continuous Blood-pressure Technology During a Total Intravenous Anaesthesia (TIVA).
Brief Title: Comparability of Invasive and Non-invasive Haemodynamic Monitoring
Acronym: HMPR1
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Tino Münster, Prof. Dr., University of Erlangen-Nürnberg Medical School
Other Study IDs: HMPR1
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Anesthesia; Anesthesia, Intravenous
Keywords: invasive arterial pressure; extended hemodynamic monitoring; propofol; remifentanil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
During general anesthesia the basic non-invasive monitoring of hemodynamic parameters (blood pressure, O2-saturation, cardiogram) is crucial. It can be enhanced to so called "extended hemodynamic monitoring" depending on the operation and patient. Frequently an invasive arterial cannula is used to provide continuous information on the blood pressure. This invasive method is very accurate and clinically established, but can be linked to adverse effects e.g. reduction of the circulation flow distal of the canulla, haematoma, infection etc. ccNexfin (Edwards Lifescience) is a finger cuff measuring the blood pressure in a non-invasive manner. It thus offers beat-to-beat information even about the extended hemodynamic parameters as cardiac output (CO), cardiac index (CI), stroke volume (SV), stroke volume index (SVI) and stroke volume variation (SSV), if connected to the clinical platform EV1000 (Edwards Lifescience).

Assuming that the two methods are equal we plan to measure extended hemodynamic parameters before, during induction and during ongoing anesthesia both invasive and non-invasive. Data will be recorded every 30sec.

Clinical evaluation of the ccNexfin technology in respect to extended hemodynamic parameters is to our knowledge rare and further assessment in this field is needed to offer patients a potentially equally reliable but less invasive monitoring. Furthermore the study should model the effect of remifentanil, propofol or its combination on haemodynamics .

ELIGIBILITY:
Inclusion Criteria:

* elective surgery with the necessity of an arterial catheter

Exclusion Criteria:

* patient not consented
* peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that get an elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | during anesthesia induction

SECONDARY OUTCOMES:
Cardiac output | during anesthesia induction
Stroke volume variation | during anaesthesia induction
Stroke volume | during anesthesia induction
Heart rate | during anaesthesia induction

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Erlangen, Bavaria, Germany